CLINICAL TRIAL: NCT04058054
Title: Skin Prick Test of KeraStat® Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KeraNetics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KSCM-CRD-002
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Results first posted 2022-09-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Histamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- KeraStat® Cream (Experimental): KeraStat® Cream is a non-sterile, non-implantable wound dressing intended to provide a moist environment in the management of a variety of partial thickness dermal wounds.
  Interventions: Device: KeraStat® Cream
- KeraStat® Gel (Experimental): KeraStat® Gel is a sterile, non-implantable water-based gelatinous (hydrogel) wound dressing intended to act as a protective covering in the management of a variety of partial thickness dermal wounds.
  Interventions: Device: KeraStat Gel
- Biafine (Experimental): Wound dressing for management of partial and full thickness wounds.
  Interventions: Device: Biafine
- Histamine (Active Comparator): Histamine is provided as a solution of histamine base (6.0 mg/mL).
  Interventions: Drug: Histamine
- Saline (Sham Comparator): Saline (sterile) is provided as a 0.9% NaCl solution.
  Interventions: Drug: Saline (0.9% NaCl)

INTERVENTIONS:
Device: KeraStat® Cream — Administered 0.025 gm of KeraStat Cream per subject on day 1 of the study.
  Arms: KeraStat® Cream
Device: KeraStat Gel — Administered 0.025 gm of KeraStat Gel per subject on day 1 of the study.
  Arms: KeraStat® Gel
Device: Biafine — Administered 0.025 gm of Biafine per subject on day 1 of the study.
  Arms: Biafine
Drug: Histamine — Administered 1 drop of Histamine Dihydrocl (6 mg/mL) per subject on day 1 of the study.
  Arms: Histamine
Drug: Saline (0.9% NaCl) — Administered 1 drop of saline per subject on day 1 of the study.
  Other Names: Sodium Chloride syringe
  Arms: Saline

SUMMARY:
To evaluate the potential for a humoral reaction to KeraStat Cream compared to a predicate device using the skin prick test.

DETAILED DESCRIPTION:
Study Overview:

Study Periods:

The length of study participation for a subject is about 2-3 days depending on availability for the final site check. There are two skin prick site checks during the course of Day 1 with a final follow up between Days 2 and 3.

Study Evaluations:

Initial screening (Screening Visit; Visit 1) will be performed on the day of the Skin Prick Test (SPT) administration and will include obtaining demographic information, brief medical history, and abbreviated physical exam.

On Day 1 (Visit 1) the SPT will be performed on the infrascapular region of the back to the right of the midline. Test articles will include the subject device (KeraStat Cream), predicate devices (KeraStat Gel, Biafine), positive control (histamine), and negative control (saline). Each test article will have a single administration, only the re-test will utilize a triplicate administration. The SPT will be ready for initial reading after approximately 15 minutes (but no sooner than 10 minutes and no longer than 20 minutes) following the final SPT administration in the series. When reading the test, the investigator will note the presence or absence of a wheal at all five sites and will measure the diameter of each wheal present. In order for the SPT to be valid, the wheal at the positive control site must exceed that at the negative control by 4 mm. If the above criteria are not met, the SPT will be repeated in triplicate on the infrascapular region of the back to the left of the midline, following the same protocol. Following the initial reading, the subject will remain at the testing facility.

A second reading will be conducted approximately 6 hours (+/- 15 minutes) after SPT administration on Day 1 (Visit 1). When reading the test, the investigator will note the presence or absence of a wheal at all five sites and will measure the diameter of each wheal present. Subjects are free to leave the clinical site after the second reading. Subjects will be instructed to promptly contact the PI and go to the ER if symptoms of an allergic reaction or shock occur.

Subjects will return to the office one to two days after initial administration for a third test reading (Visit 2). When reading the test, the investigator will note the presence or absence of a wheal in all five sites and will measure the diameter of each wheal present. Each site of test article administration will be measured for a positive reaction. A positive reaction is present when there is a measurable wheal of 3 mm or more, surrounded by a flare. Small wheals are to be confirmed by palpation. A flare alone is disregarded.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 18-65
2. Able to understand the informed consent and provide written informed consent
3. Healthy, unmarked skin at the test area
4. Agreement to avoid consumption of antihistamines until completion of third test reading (Visit 2)

Exclusion Criteria:

1. Women who are pregnant, lactating/nursing or plan to become pregnant
2. Presence of skin disease, such as widespread urticaria or eczema
3. Diagnosis of infectious disease
4. Receiving corticosteroids, immunosuppressive agents, radiation or chemotherapy, topical growth factors, anxiolytics, imipramine, phenothiazine, dopamine, phenergen, clonidine, montelukast, immunotherapy, UV light therapy, H-2 antagonist, cyclosporine or any other medication the investigator feels will affect the test within the last month
5. Medical history of hypotension, severe hypertension, vasomotor instability, asthma, autoimmune disease, severe cardiac, pulmonary or renal disease
6. Tattoo in the intrascapular test area
7. History of surgical procedure/skin graft in the intrascapular test area
8. Employee or relative of employee of KeraNetics
9. Consumption of an anti-histamine within 7 days of the screening visit
10. History of hypersensitivity to histamine products
11. Any condition the investigator determines will compromise subject safety or prevent the subject from completing the study
12. Participated in an investigational study within 30 days of the screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Wilson, DO, Principal Investigator — PMG Research
Locations (1):
- PMG Research, Inc., Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Skin prick site
Period: Overall Study
Arm/Group | KeraStat® Cream | KeraStat® Gel | Biafine | Histamine | Saline
Started | 22; 22 Skin prick site | 22; 22 Skin prick site | 22; 22 Skin prick site | 22; 22 Skin prick site | 22; 22 Skin prick site
Completed | 22; 22 Skin prick site | 22; 22 Skin prick site | 22; 22 Skin prick site | 22; 22 Skin prick site | 22; 22 Skin prick site
Not Completed | 0; 0 Skin prick site | 0; 0 Skin prick site | 0; 0 Skin prick site | 0; 0 Skin prick site | 0; 0 Skin prick site

BASELINE CHARACTERISTICS:
Groups:
- Main Study Group: This study utilized intrasubject comparisons, so each subject received each treatment.
Arm/Group | Main Study Group
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Reaction to Test Article
Description: Wheal measurement in millimeters (mm)
Time Frame: assessed at 15 min, 6 hours, 24-48 hours; 15 min reported
Population: each unique treatment was applied to a single prick lesion on each participant's back
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: skin pricks
Arm/Group | KeraStat® Cream | KeraStat® Gel | Biafine | Histamine | Saline
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
Number analyzed (skin pricks) | 22 | 22 | 22 | 22 | 22
mm | 0 (0) | 0.32 (1.49) | 0.23 (1.07) | 6.73 (0.34) | 0 (0)

ADVERSE EVENTS:
Time Frame: two days
Groups:
- Main Study Group - KeraStat Cream: KeraStat® Cream is a non-sterile, non-implantable wound dressing intended to provide a moist environment in the management of a variety of partial thickness dermal wounds. Administered 0.025 gm of KeraStat Cream per subject on day 1 of the study.
- Main Study Group - KeraStat Gel: KeraStat® Gel is a sterile, non-implantable water-based gelatinous (hydrogel) wound dressing intended to act as a protective covering in the management of a variety of partial thickness dermal wounds. Administered 0.025 gm of KeraStat Gel per subject on day 1 of the study.
- Main Study Group - Biafine: Wound dressing for management of partial and full thickness wounds. Administered 0.025 gm of Biafine per subject on day 1 of the study.
- Main Study Group - Histamine: Histamine is provided as a solution of histamine base (6.0 mg/mL). Administered 1 drop of Histamine Dihydrocl (6 mg/mL) per subject on day 1 of the study.
- Main Study Group - Saline: Saline (sterile) is provided as a 0.9% NaCI solution. Administered 1 drop of saline per subject on day 1 of the study.
  Other Names:
  Sodium Chloride syringe
Arm/Group | Main Study Group - KeraStat Cream | Main Study Group - KeraStat Gel | Main Study Group - Biafine | Main Study Group - Histamine | Main Study Group - Saline
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT04058054/Prot_SAP_000.pdf